CLINICAL TRIAL: NCT07226336
Title: Testing a Dissonance-Based Intervention to Reduce Ultra-Processed Food Consumption Via Activism Against the Food Industry
Brief Title: Dietary Interventions to Reduce Ultra-Processed Food Intake
Acronym: DISRUPT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Charlotte Hagerman, Principal Investigator, Research Scientist, Oregon Research Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 31272E; 5P30DK111022 (NIH)
Record Dates: First submitted 2025-10-31; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Ultra-Processed Food Intake; Obesity & Overweight
Keywords: Ultra-Processed Food; Dietary Change; Cognitive Dissonance
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Control Condition (Active Comparator): Participants in this condition (Standard Dietary Change OFF, Dissonance OFF) will receive an educational workshop on UPFs and their harmful health effects.
  Interventions: Behavioral: Introductory Educational Workshop
- Standard Dietary Change Strategies (Experimental): Participants in this condition (Standard Dietary Change ON, Dissonance OFF) will attend an introductory educational workshop about UPFs, then attend weekly group sessions that teach standard dietary change strategies for the next 7 weeks.
  Interventions: Behavioral: Introductory Educational Workshop; Behavioral: Standard Dietary Change (ON/OFF)
- Dissonance Strategies (Experimental): Participants in this condition (Standard Dietary Change OFF, Dissonance ON) will attend an introductory educational session about UPFs, then attend weekly group sessions in which they will be engaged in cognitive dissonance-inducing activities for the next 7 weeks.
  Interventions: Behavioral: Introductory Educational Workshop; Behavioral: Cognitive Dissonance Strategies (ON/OFF)
- Standard Dietary Change+ Dissonance Strategies (Experimental): Participants in this condition (Standard Dietary Change ON, Dissonance ON) will attend an introductory educational session about UPFs, then attend weekly group sessions in which they will 1) learn standard dietary change strategies and 2) be engaged in cognitive-dissonance inducing strategies for the next 7 weeks. Groups will be slightly longer to accommodate both intervention strategies.
  Interventions: Behavioral: Introductory Educational Workshop; Behavioral: Standard Dietary Change (ON/OFF); Behavioral: Cognitive Dissonance Strategies (ON/OFF)

INTERVENTIONS:
Behavioral: Introductory Educational Workshop — Participants will attend an introductory educational workshop held through videoconferencing software in week 1 of the program. The workshop will teach participants about ultra-processed foods (UPFs) and their negative health effects.
Behavioral: Standard Dietary Change (ON/OFF) — Participants randomly assigned to have Standard Dietary Change Strategies ON will attend group sessions with a study coach, during which they will learn standard dietary change strategies such as meal planning, problem solving, and goal setting. Sessions will involve didactics, discussion, and interactive elements to promote greater participant engagement.
  Arms: Standard Dietary Change Strategies; Standard Dietary Change+ Dissonance Strategies
Behavioral: Cognitive Dissonance Strategies (ON/OFF) — Participants assigned to have the dissonance condition ON will attend weekly virtual group sessions with a coach, during which they will learn about the nefarious efforts of the food industry, including its creation of UPFs to be hyperpalatable and addictive, its predatory and deceptive marketing techniques, and its role in blocking policy change. Special emphasis will be placed on the food industry's exploitation of vulnerable, low-income communities by inundating these neighborhoods with cheap, ultra-rewarding products. Participants will be asked to engage in activities designed to elicit cognitive dissonance for consuming UPFs. Examples include writing letters to Congress urging policy change and creating "elevator pitches" for family and friends.
  Arms: Dissonance Strategies; Standard Dietary Change+ Dissonance Strategies

SUMMARY:
The DISRUPT clinical trial will test two different 2-month programs to help adults with overweight/obesity (N=60) reduce their intake of ultra-processed foods (UPFs). Participants will be randomly assigned to receive standard dietary change strategies, cognitive dissonance strategies that engage them in activism against the UPF industry, or both. All participants will attend an introductory educational workshop about UPFs. If they are assigned to receive one or more of these strategies, they will attend weekly group sessions with the relevant intervention content for 7 more weeks. Groups will be held virtually.

DETAILED DESCRIPTION:
The DISRUPT clinical trial will test 2-month interventions for reducing ultra processed food (UPF) intake among 60 adults with overweight or obesity (ages 18-70) who frequently consume UPFs. Participants will be randomly assigned to receive a standard dietary change (SDC) intervention (ON/OFF), in which they will receive the typical toolbox of evidence-based methods for changing diet (e.g., meal planning, problem solving, reflecting on the benefits of change) to help them reduce their ultra-processed food intake. Participants will be also randomly assigned to receive a cognitive dissonance intervention (ON/OFF). In this intervention, participants will learn about the harms of the food industry and be engaged in activism against this industry to elicit cognitive dissonance for consuming UPFs. Participants will be randomly assigned to each condition separately (through a 2x2 factorial design, resulting in four possible experimental conditions: 1) Control (both OFF), 2) Standard Dietary Change Condition (SDC ON, Dissonance OFF), 3) Dissonance Condition (SDC OFF, Dissonance ON), and 4) SDC + Dissonance Condition (SDC ON, Dissonance ON).

All participants will receive an introductory educational workshop on UPFs, how to identify them, and their harmful health effects. Participants assigned to receive at least one of the interventions (i.e., SDC, dissonance, or both) will attend weekly group sessions for weeks 2-8.

Aim 1 is to test the isolated and interactive effects of standard behavior change strategies and dissonance-based strategies on treatment outcomes. Participants randomly assigned to the SDC condition and the Dissonance condition, respectively, are expected to have larger reductions in UPF intake, greater improvements in indicators of dietary quality (e.g., added sugar, sodium intake), and more weight loss, compared to those in the control condition. The effect of the SDC + Dissonance condition (vs. the control condition) on treatment outcomes is expected to be synergistic, greater than the additive effect either condition alone.

Aim 2 is to test the hypothesis that having the dissonance intervention ON will attenuate the disparity in treatment outcomes for individuals with socio-structural barriers to healthy eating (i.e., low perceived socioeconomic status, low income, limited access to healthy food, and unhealthy neighborhood food environment).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 years old
* BMI >25 and <50 kg/m2
* Wish to reduce their UPF intake
* Consume at least 2 UPF items per day and at least 4 distinct UPF items per week

Exclusion Criteria:

* Have ever been diagnosed with anorexia nervosa or bulimia nervosa
* Are using medications known to influence eating behavior and/or weight (e.g., semaglutide)
* Currently using insulin
* History of bariatric surgery
* Current pregnancy or planning to become pregnant during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Ultra-Processed Food Intake | Baseline, Post-Treatment (2 months)
  Dietary intake will be assessed using the Automated Self-Administered 24-hour Dietary Recall (ASA24), in which participants report all of the food and beverages consumed during the past 24 hours. At each assessment, participants will complete three recalls (two weekdays, one weekend day). To calculate UPF intake, each food entry on the ASA24 will be coded into a NOVA category based on a classification system developed through a collaboration between The University de São Paulo and the National Cancer Institute. UPF intake will be operationalized as the average daily calories that come from UPFs.

SECONDARY OUTCOMES:
Weight | Baseline, Post-Treatment (2 months)
  Participants will be asked to provide their current weight by weighing themselves on three consecutive mornings on a digital scale following proper weighing procedures (e.g., in the morning, in a fasted state). The average of the three days of weights will be used.
Added Sugar Intake | Baseline, Post-Treatment (2 months)
  Average daily added sugar intake (in grams) will be generated from participants' ASA24 recalls.
Saturated Fat Intake | Baseline; Post-Treatment (2 months)
  Average daily saturated fat intake (in grams) will be generated from participants' ASA24 recalls.
Sodium Intake | Baseline; Post-Treatment (2 months)
  Average daily sodium intake (in milligrams) will be generated from participants' ASA24 recalls.
Fruit Intake | Baseline; Post-Treatment (2 months)
  Average daily fruit intake (in cups) will be generated from participants' ASA24 recalls.
Vegetable Intake | Baseline; Post-Treatment (2 months)
  Average daily vegetable intake (in cups) will be generated from participants' ASA24 recalls.
Total Calorie Intake | Baseline; Post-Treatment (2 months)
  Average daily calorie intake will be generated from participants' ASA24 recalls.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Hagerman, PhD, Principal Investigator — Oregon Research Institute

IPD SHARING:
Plan to Share IPD: Yes
Identifiable data will be de-identified prior to submission in the public repository to protect research participant privacy and confidentiality. All individual-participant level data will be preserved and shared, as all variables collected are pertinent to scientific questions.
Supporting Information: Analytic Code
Time Frame: IDP and supporting information will be shared within 12 months of the trial's completion, and will be stored indefinitely.